CLINICAL TRIAL: NCT02327832
Title: Safety Study of a Less Invasive Liver Regeneration Therapy Using Cultured Autologous Bone Marrow-derived Mesenchymal Stem Cells for Compensated Liver Cirrhotic Patient
Brief Title: Safety Study of Liver Regeneration Therapy Using Cultured Autologous BMSCs
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yamaguchi University Hospital (Other)
Responsible Party: Principal Investigator, tarotakami, MD, PhD, Yamaguchi University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICHINAI-BMSC1
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Liver Regeneration
Keywords: Confirmation; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous BMSCs (Experimental): Infusion of cultured autologous bone marrow derived mesenchymal stem cells
  Interventions: Procedure: Autologous BMSCs; Drug: bone marrow-derived mesenchymal stem cells

INTERVENTIONS:
Procedure: Autologous BMSCs — Cultured autologous bone marrow-derived mesenchymal stem cells
  Other Names: BMSC
Drug: bone marrow-derived mesenchymal stem cells

SUMMARY:
Patients eligible for this study include those with decompensated liver cirrhosis with a Child-Pugh score ≥7 (Child-Pugh B) in whom further improvement with current medical treatment is not expected. Other inclusion criteria are age 20 to 75 years and a serum total bilirubin of 3.0 to 5.0 mg/dL, or if the total bilirubin is <3.0 mg/dL, patients who are still deemed unsuitable as a candidate for general anesthesia. About 30 mL of autologous bone marrow was collected from the bilateral iliac crests under local anesthesia, heparin was added after collection. In addition, at the Center for Regenerative and Cell Therapy at Yamaguchi University Hospital, a nucleated cell fraction was prepared. Next, a cell suspension was prepared by adding culture medium, and this was inoculated into a culture flask. After subculturing for 3 weeks, the cells were infused through a peripheral vein. The primary endpoint is the incidence of adverse events up to 24 weeks after ABMSC infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for this study include those with decompensated liver cirrhosis with a Child-Pugh score ≥7 (Child-Pugh B) in whom further improvement with current medical treatment is not expected. Other inclusion criteria are age 20 to 75 years and a serum total bilirubin of 3.0 to 5.0 mg/dL, or if the total bilirubin is <3.0 mg/dL,
* Patients who are still deemed unsuitable as a candidate for general anesthesia.
* Patients must provide informed consent for study participation.

Exclusion Criteria:

* Patients with a current history of malignant neoplasm.
* Patients with gastroesophageal varices at risk of rupture.
* Patients with renal insufficiency and a serum creatinine ≥2 mg/dL.
* Patients with a hemoglobin <8 g/dL, a platelet count <50,000/μL, or a prothrombin time <40%.
* Patients with a performance status of 3 or 4.
* Patients who refuse to consent to allogeneic blood transfusion.
* Women who are pregnant.
* Patients whom their attending physician deems are not suitable candidates for general anesthesia.
* Patients with a current or previous severe allergic reaction to a contrast agent, beef, cow milk, and anesthesia.
* Any patient deemed unsuitable for study inclusion by their attending physician.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events | up to 24 weeks the infusion

SECONDARY OUTCOMES:
Child-Pugh score | up to 24 weeks the infusion
Serum albumin levels | up to 24 weeks the infusion
Serum fibrosis markers | up to 24 weeks the infusion
Improvement or disappearance of lower extremity edema | up to 24 weeks the infusion
Subjective symptom scores (SF-36) | up to 24 weeks the infusion

CONTACTS AND LOCATIONS:
Overall Officials: Isao Sakaida, MD, PhD, Study Chair — Yamaguchi University Hospital
Locations (1):
- Department of Gastroenterology and Hepatology Yamaguchi University Graduate School of Medicine, Ube, Yamaguchi, Yamaguchi, Japan